CLINICAL TRIAL: NCT00447720
Title: Translation of CDC and NIDA Programs to Prevent HIV/AIDS Among Persons With Serious Mental Illness
Brief Title: HIV Prevention Among Substance Abusing SMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael Blank, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 704260; 5R01DA015627-03 (NIH)
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Mentally Ill Persons; Substance Abuse; HIV Infections
Keywords: HIV prevention skills; Seriously Mentally Ill (SMI); Substance abuse; Philadelphia; HIV seronegativity
MeSH Terms: conditions — Substance-Related Disorders; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PATH counseling (Experimental): These participants received the PATH intervention
  Interventions: Behavioral: PATH
- Treatment as Usual (Active Comparator): These individuals receive treatment as they normally would receive in the community
  Interventions: Behavioral: PATH

INTERVENTIONS:
Behavioral: PATH — We have chosen to translate two proven prevention programs for delivery to the SMI populations by their case managers. These interventions are the Brief Counseling intervention from the Project Respect program and the Community-Based Outreach Program (CBOM). Together we will translate them into ongoing case management for SMI persons who also abuse substances in the Preventing AIDS through Health Project (PATH). Consistent with other findings regarding HIV infections among the SMI, in our preliminary studies we found that these individuals are at much higher risk within the population of persons being served in Philadelphia.

SUMMARY:
This study seeks to examine the effectiveness of translating two proven interventions, RESPECT, and the NIDA Community Based Outreach Model, into one program of education, PATH, to be delivered by case managers to their seriously mentally ill, substance abusing clients.

The objective is to teach case managers to assess the specific risk profiles of their clients, and then create a plan of intervention aimed at reducing high risk sexual and substance abusing behaviors.

DETAILED DESCRIPTION:
Persons with serious mental illness (SMI) are at increased risk for HIV/AIDS. The relative risk of HIV/AIDS is at least five times greater in SMI as the general Medicaid population in Philadelphia and over seven times for those also treated for substance abuse. We will implement a prevention program for persons with SMI who also abuse substances over five years at a local Community Mental Health Center. Preventing AIDS Through Health (PATH) is a translation of two HIV prevention programs proven effective in the general population and among substance users. Both are highly structured, manualized interventions. PATH uses mental health case managers to draw on features of both interventions depending on individual consumer risk profiles. These case managers have special expertise in providing services to this population and we believe that this expertise, prior relationships with these persons, and an ability to regularly reinforce the intervention will result in significantly reduced risk. There are two sets of research participants - the persons with SMI as well as the case managers themselves. Informed consent will be obtained from both sets of participants.

It is estimated that approximately 300 individuals with mental illnesses will participate; with 150 assigned to the control group and 150 assigned to the treatment group. There will be approximately 32 participating case managers whose caseloads will be randomized to treatment.

Blood testing will identify those who are HIV positive at baseline. Breathalyzer and urine testing will supplement clinical interviews and other measures to identify substance abuse co-morbidity. Using a longitudinal experimental and control group design, we will randomly assign case managers to deliver the intervention to consenting participants in their caseloads who meet inclusion criteria. Independent interviews will be conducted with case managers before the intervention, and again at 3,6,and 12-months post intervention and focus on changes in risk behaviors, fidelity of translation of the intervention, cost and outcomes. Breathalyzer and urine tests at 12-months will supplement self-reports of use of alcohol, cocaine, marijuana, benzodiazepines, and opiates.

This is minimal risk research. The potential exists for great benefits to the mental health system at large. Potential risks are quite reasonable given the safeguards proposed and the valuable information to be yielded on the development of responsive interventions and practices to improve care for urban SMI who are at risk for HIV infection. The potential risks for participants in the study are not expected to be greater than those obtained during the performance of routine psychological or physical examinations or tests. All instruments used in primary data collection are those that are frequently used in similar research with similar populations and have not been associated with any adverse events. The questions that will be asked of the research participant pose no more risk than those they would respond to in the course of treatment. That is, the questions are similar to those that mental health professionals ask in the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of case management at Hall Mercer Community Health Center
* Use of substance or history of using substances
* Sexual activity or interest in a sexual relationship sometime in the future

Exclusion Criteria:

* May not be HIV+

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2004-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Outcome measures used for calculating effectiveness will be reduction in sexual and substance-use-related risk behaviors. Other outcomes include improved condom use as well as increase in knowledge of HIV. | 24 months
Condom skills | baseline, 6,12
  Behavioral skills

SECONDARY OUTCOMES:
Behavioral risk self report | baseline, 6, 12, and 24 months
HIV risk reduction | baseline, 6, 12 months
  Self-report

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blank, PhD, Principal Investigator — Center for Mental Health Policy and Services Research
Locations (1):
- Hall Mercer Community Mental Health Clinic, Philadelphia, Pennsylvania, United States